CLINICAL TRIAL: NCT05065593
Title: The Effect of Aerobic and Resistant Exercise Training on Hepatic Functions, Inflammatory Markers and Functional Capacity in Patients With Non-Alcoholic Steatohepatitis
Brief Title: The Effect of Aerobic and Resistant Exercise Training in Patients With Non-Alcoholic Steatohepatitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Birgul Kumbaroglu, Research Assistant, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA- 21027
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: fibrosis; exercise; inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face Training Group (Experimental): After completing all assessments, the intervention group will participate in face-to-face exercise training with a physiotherapist for 3 days for 4 months.
  In the first week, patients will be taught body awareness; parameters of correct loading on the muscle will be explained and the limits of safe exercise will be drawn. At the beginning and end of all exercises, there will be short-term active stretching and relaxation exercises performed by the patient as a warm-up and cool-down period. In the first 4 weeks, it is planned to increase the physical fitness levels of individuals with progressive resistance exercises and to make them suitable for aerobic loading. For each patient, the PRE, resistance will be increased from 60% to 80% for as long as the person can. At the end of the 1st month, the time allocated to resistance exercise training will be reduced and until the end of the 4th month, an increasing intensity aerobic exercise training will be given on the stationary bike.
  Interventions: Other: resistance and aerobic exercise
- Home-Based Control Group (Active Comparator): After the patients assigned to the control group are evaluated by the physiotherapist with field tests and scales for physical functions, the patients will be informed about the importance of lifestyle changes in disease management, gait training will be given to increase their physical activity level and participants will be asked to follow a 45-minute walking program every day within their own means. All patients in the control group will be followed up regularly and their activity levels will be questioned in interim evaluations by asking them to keep a weekly physical activity diary.
  Interventions: Other: physical activity recommendation

INTERVENTIONS:
Other: resistance and aerobic exercise — Resistive exercises allow loading the muscle under suitable conditions with various weights or resistances. In order to increase the level of physical fitness with the increase of muscle strength and bone mass in individuals, resistance exercises were preferred. Aerobic exercises, on the other hand, are a special type of exercise that develops both the musculoskeletal system and the cardiovascular system, which includes large muscle groups and should be performed for at least 20 minutes when the heart rate accelerates at certain rates. Aerobic exercise was preferred in order to increase cardiovascular endurance, accelerate fat burning and reduce fatigue.
  Arms: Face-to-Face Training Group
Other: physical activity recommendation — Patients will be informed about the importance of lifestyle change in disease management, walking training will be given to increase their physical activity level, and participants will be asked to follow a 45-minute walking program every day within their own means.
  Arms: Home-Based Control Group

SUMMARY:
The term non-alcoholic fatty liver disease (NAFLD) is used to describe a range of chronic liver diseases that range from steatosis to steatohepatitis, advanced fibrosis, cirrhosis, or excessive alcohol consumption or other causes of steatosis. In this spectrum, Non-Alcoholic Steatohepatitis (NASH), which defines liver damage accompanied by steatosis and inflammation (hepatitis), is one of the most common causes of chronic liver disease worldwide, especially in developed and developing countries, and is present in 15-35% of the general population. Individuals diagnosed with NASH primarily experience deterioration in liver functions, but patients are also affected in terms of vascular structures, immunopathological responses, functional and psychosocial conditions. It is seen that in addition to intrahepatic lipid content, inflammatory markers, liver enzymes, and liver functions, cardiopulmonary endurance, physical activity level, and muscle strength are also affected in these patients, so it is evaluated for the diagnosis and planning of the treatment of the disease. There is no drug with proven efficacy in the treatment of the disease. Since a significant proportion of NASH patients have obesity, Type II Diabetes Mellitus or dyslipidemia, the focus of treatment is to control risk factors or protect the liver from harmful factors such as TNFα. Therefore, the mainstay of treatment, for now, seems to be weight control with a lifestyle change, including regular exercise training and diet control. Exercise intervention is considered an essential component of NAFLD treatment, however; there are a limited number of published articles showing the effects of exercise training in the management of NASH. In addition, the physiological effect of exercise has still not been clarified because NASH is accompanied by metabolic problems such as obesity and T2DM. This study, it is aimed to bring innovation to the literature in understanding the physiological effects of exercise for this disease group by examining the effects of resistance exercise training in addition to aerobic exercise on intrahepatic lipid content, liver functions, inflammatory markers, muscle strength, functionality, and biopsychosocial status in individuals with NASH diagnosis who do not have an additional metabolic problem.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with NASH according to the diagnostic criteria determined by the American Gastroenterology Society / Asia-Pacific Working Group,
* No history of hepatic decompensation such as hepatic encephalopathy or abdominal ascites,
* Not being obese according to the criteria of the World Health Organization (Body Mass Index (BMI) <30),
* HbA1c value <6.5%,
* No changes in blood pressure, hyperlipidemia drugs in the last 3 months,
* Absence of any mental disorder or exercise compliance problem that would prevent them from participating in the study.
* It was determined as being voluntary to participate in the study.

Exclusion Criteria:

* A history of liver disease other than NASH, such as acute or chronic viral hepatitis, autoimmune hepatitis,
* Alcohol consumption >30 g/day in men and >20 g/day in women,
* Having regular exercise habits,
* Presence of conditions where exercise is contraindicated, such as unstable ischemia, decompensated heart failure, arrhythmia that increases with exercise and cannot be controlled, severe aortic stenosis, hypertrophic cardiomyopathy,
* Having orthopedic problems that limit lower extremity movements such as previous cerebrovascular disease, neurological diseases that cause cognitive and motor loss such as Alzheimer's and Parkinson's, and endoprosthesis surgery in the last three months, permanent joint contracture,
* Regular use of food supplements,
* It was determined that he did not volunteer to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline intrahepatic lipid percentage | Change from baseline intrahepatic lipid percentage to 16th week
  Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) is a MRI-based diagnostic imaging biomarker of the liver, developed in order to facilitate, by enriching, patient recruitment for clinical trials in NASH. The PDFF method is the most objective method for lipid measurement in the liver.
Change from baseline hepatic steatosis percentage | Change from baseline steatosis percentage to 16th week
  Magnetic Resonance Elastography (MRE) is a technology that combines MRI imaging with low-frequency vibrations to create a visual map (elastogram) that shows the stiffness of body tissues. Currently, MRE is used to detect stiffening of the liver caused by fibrosis and inflammation in chronic liver disease. In chronic liver disease, before reaching the stage of cirrhosis, while detecting fibrosis in the early stages, a tissue stiffness map called elastogram can be drawn. Because the waves can be visualized and analyzed deep in the liver, MRE can evaluate much larger amounts of the total liver than a liver biopsy and has been shown to have high diagnostic accuracy in studies.
Change of liver function parameters level | Change from baseline liver function parameters level to 16th week
  Routine liver function test results including alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), albumin, and bilirubin will be measured. All parameters will be recorded in IU/L.The ALT and AST tests measure enzymes that the liver releases in response to damage or disease. The albumin test measures how well the liver creates albumin, while the bilirubin test measures how well it disposes of bilirubin. ALP can be used to evaluate the bile duct system of the liver.
Change of lipid panel | Change from baseline lipid panel values to 16th week
  The lipid panel analysis contains total cholesterol, Low-density lipoprotein (LDL) cholesterol, High-density lipoprotein (HDL) cholesterol, triglycerides. All parameters will be recorded in mg/dL. Higher than normal cholesterol levels are associated with cardiovascular and metabolic diseases. Also, high total cholesterol LDL or triglyceride ratios are associated with NASH. Therefore, the lipid profile is evaluated to monitor NASH progression.

SECONDARY OUTCOMES:
Evaluation of inflammatory markers | 5 minutes, through study completion, an average of 16 weeks, change from baseline inflammatory marker status at 16 weeks.
  At the beginning of the study and at the end of the 4th month corresponding to the end of the treatment, the cytokine serum levels of all individuals will be measured by the specialist physician. These cytokines; The proinflammatory cytokine hsCRP, TNF α, which is one of the primary indicators of inflammation, has been determined as IL-6, which gives the earliest and most effective response to exercise and has an anti-inflammatory effect when released from the muscle, IL-10, which is an anti-inflammatory cytokine, and TGF β, which plays a central role in liver fibrogenesis. For measurement, 10 ml of blood sample for each cytokine will be taken from each patient, and the serum will be separated into a dry tube and stored frozen for further blood analysis at -20 °C until measurement.
Evaluation of aerobic capacity | 12 minutes, through study completion, an average of 16 weeks, change from baseline aerobic capacity at 16 weeks.
  Maximum Oxygen Consumption (VO2max) measurement is accepted as an easy, reliable and best indicator of aerobic capacity. Although a direct measuring device was considered for the study, considering the pandemic due to Covid-19, it was thought that even if it was disinfected for each patient, it would pose a risk due to contamination in the face mask of the device and the pipes that provide the air flow to the device. For this reason, aerobic capacity will be evaluated with the Increasing Speed Shuttle Walk Test (ISWT), which is one of the indirect measurement methods. This test is an exercise test in which walking between two cones 10 m apart at increasing speed for 12 minutes is counted as one sit-up for each 10-meter walk between the two cones. It is continued until the patient is unable to continue the test due to shortness of breath, the heart rate reaches 85% of the maximum expected heart rate, or completes the 12-minute test.
Evaluation of physical activity level | 5 minutes, through study completion, an average of 16 weeks, change from baseline physical activity level at 16 weeks.
  It will be done with the International Physical Activity Questionnaire-Short Form (IPAQ-SF). There are eight versions of the questionnaire in total, but the short form "last 7 days" will be used in this study. The short form (7 questions) provides information about the time spent in walking, moderate-to-vigorous and vigorous activities. The time spent sitting is considered a separate question. It is classified as low, medium, and high level by calculating the activity level of the person in terms of METs according to the duration, frequency, and intensity level of the movement. The Turkish version study was done by Sağlam et al.
Evaluation of muscle strength | 10 minutes, through study completion, an average of 16 weeks, change from baseline fatique status at 16 weeks
  "Nicholas Manual Muscle Tester (Model 01165, Lafayette Instrument Company, Lafayette, Indiana, USA)" will be used for an objective evaluation. Since training will be given for large group muscles, muscle strength of hip, knee, shoulder and elbow flexors and extensors will be evaluated. The position of the dynamometer will be standardized for each measurement. The standard instruction, "push as hard as you can", will be given to the subject for each trial by applying a constant resistance for 3 to 5 seconds, directed perpendicular to the long axis of the measured extremity, in the test device to induce isometric muscle contraction. 3 repetitions will be done for each muscle group and the highest score will be recorded in kilograms (kg).
Evaluation of fatigue | 5 minutes, through study completion, an average of 16 weeks, change from baseline fatique status at 16 weeks
  The Fatigue Severity Scale (FSS) will be used, the Turkish validity and reliability study of which was conducted by Armutlu et al. It is a self-report scale consisting of 9 items that evaluates the degree of fatigue severity in the last 1 week. According to a 7-point Likert scale for each item, the most appropriate one of the statements ranging from 7=strongly agree to 1=strongly disagree is marked by the patient. The scores obtained from each item are added together and the total value is divided by 9. 4.0 is used as the cut-off value for fatigue in studies.
Evaluation of pain | 5 minutes, through study completion, an average of 16 weeks, change from baseline pain status at 16 weeks
  The presence of pain of the participants will be questioned; If there is pain, it will be requested to be marked on the body diagram and its duration, localization, frequency, triggering factors, and whether it occurs during rest and activity will be recorded. In addition, using the Visual Analogue Scale (VAS), the patient will be asked to mark the severity of the pain on a 10-centimeter line, and it will be measured with a ruler and recorded out of 10. Pain intensity can take the lowest 0 and the highest 10 value. A higher score means worsening of pain.
Evaluation of quality of life | 10 minutes, through study completion, an average of 16 weeks, change from baseline quality of life at 16 weeks
  ts validity and reliability have been established in healthy individuals and in various disease groups, and the quality of life will be evaluated with the Short Form-36 (SF-36), the first Turkish validity and reliability of which was made by Koçyiğit et al. (46). General health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons and vitality are 8 sub-parameters of SF-36 and it includes 11 questions consisting of 36 items. Each sub-parameter is scored between 0 and 100 points, and a high score indicates good health.
Evaluation of anxiety and depression | 7 minutes, through study completion, an average of 16 weeks, change from baseline anxiety and depression status at 16 weeks
  The Hospital Anxiety and Depression Scale (HADS) was developed to identify possible cases of anxiety disorder and depression in hospital clinics. The scope of use of the scale is not for diagnostic purposes, but to reveal depression and anxiety accompanying existing diseases. Turkish validity and reliability were performed by Aydemir et al. It is a 14-item scale consisting of the Anxiety subscale (HADS-A) and the Depression subscale (HADS-D), both of which contain seven items. The answer to each question is scored between 0-3 using a four-point Likert scale, and both sub-parameters can take a value between 0 and 21. Scores between 0 and 7 for each of the anxiety and depression parameters are considered "normal"; A score of 8 to 10 is considered a "probable case" and a score of 11 to 21 is considered a "probable case of anxiety/depression". These cutoff points were validated with a sensitivity and specificity of around 0.80 to clinical interviews.
Evaluation of dynamic balance | 5 minutes, through study completion, an average of 16 weeks, change from baseline dynamic balance at 16 weeks
  The Timed Up and Go Test (TUG) will be used to evaluate balance and determine the risk of falling. The TUG test is an easy-to-use field test that has proven validity and reliability, and provides information about the dynamic balance of individuals and the risk of falling. For this test, the subject will be asked to get up from an armless chair and walk three meters, then turn around and sit down again. The elapsed time will be noted, the test will be repeated 3 times and the average time will be calculated.
Evaluation of body mass index (BMI) | 5 minutes, through study completion, an average of 16 weeks, change from baseline body mass index at 16 weeks
  The height of the individuals will be measured with a Dikomsan brand stadiometer with the head in the Frankfort plane and the feet closed. Bodyweight (kg), body fat amount (kg), and lean body weight (kg) will be measured with Tanita BC 780 model body analyzer. Weight and height will be combined to report BMI in kg/m^2
Evaluation of body fat percentage | 5 minutes, through study completion, an average of 16 weeks, change from baseline body fat percentage at 16 weeks
  Body fat percentage (%), and lean body weight ratio (%) will be measured with Tanita BC 780 model body analyzer.
Daily calorie follow-up | 5 minutes, through study completion, an average of 16 weeks, change from baseline daily diet statusat 16 weeks
  The patients will be given a Low-Fat Diet Program, which is a routine nutritional treatment, at the first meeting. The food consumption records of the patients will be taken with a 24-hour retrospective reminder method during the dietitian visits. Food consumption records will be evaluated using the Nutrition Information Systems (BeBiS) Package Program.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)